CLINICAL TRIAL: NCT05891275
Title: Characterization of Patients With Geographic Atrophy (GA) in the US
Brief Title: Patients With Geographic Atrophy and Their Patient Journey in the United States (US)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1484-0014
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a Geographic Atrophy diagnosis: Patients diagnosed with geographic atrophy (GA) in at least one eye, at least 50 years old with information on laterality, and registered in the Vestrum health database between January 2015 and April 2023.

SUMMARY:
To quantify and describe patients with a Geographic Atrophy (GA) diagnosis in at least one eye, and the progression to neovascular Age-Related Macular Degeneration (including how many receive Anti-VEGF), or to GA (in the fellow eye only).

ELIGIBILITY:
Inclusion Criteria:

- All patients ≥50 years, with a GA diagnosis in at least one eye, included in the Vestrum database identified during the study period (January 2015 to April 2023).

Exclusion Criteria:

- Patients without the information of laterality will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US patients ≥50 years, with a Geographic Atrophy diagnosis in at least one eye
Sampling Method: Non-Probability Sample
Enrollment: 68563 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas HQ, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational cohort study based on existing data aimed to quantify and describe patients with a diagnosis of geographic atrophy (GA) in at least one eye, the progression to wet or neovascular age-related macular degeneration (wAMD) in both eyes, and the progression to GA in the fellow eye.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included. Subjects from the Vestrum database aged 50+ with information on laterality, and a GA diagnosis between January 1, 2015, to April 30, 2023, were analyzed. While both eyes participated in the study, one eye per participant was analyzed for outcome measures.
Groups:
- Patients With Geographic Atrophy (GA): Patients diagnosed with geographic atrophy (GA) in at least one eye, at least 50 years old with information on laterality, and registered in the Vestrum health database between January 2015 and April 2023.
Period: Overall Study
Arm/Group | Patients With Geographic Atrophy (GA)
Started | 68563
Completed (Completed includes all subjects who contributed at least a data point to the analysis.) | 68563
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients diagnosed with geographic atrophy (GA) in at least one eye, at least 50 years old, with information on laterality and registered in the Vestrum health database between January 2015 and April 2023.
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 68563
Age, Continuous [Mean (Standard Deviation); unit: Years] | 82 (9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 44046
  Male | 23632
  Not specified | 885
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
GA laterality [Count of Participants; unit: Participants] — Data on the number of participants with information on laterality and registered in the Vestrum health database between January 2015 and April 2023 is presented. Only participants with available data were included in the analysis.
  Participants
    Participants with unilateral GA | 36221
    Participants with bilateral GA | 32342
Wet (neovascular) age-related macular degeneration (wAMD) [Count of Participants; unit: Participants] — Data on the number of participants with information on wet (neovascular) age-related macular degeneration and registered in the Vestrum health database between January 2015 and April 2023 is presented. Only participants with available data were included in the analysis.
  Participants
    Study eye with wAMD | 12937
    Study eye without wAMD | 55626
    Fellow eye with wAMD | 28728
    Fellow eye without wAMD | 39835
Lesion location at index [Count of Participants; unit: Participants] — Data on the number of participants with information on location of lesion at index in the study eye, and registered in the Vestrum health database between January 2015 and April 2023 is presented. Only participants with available data were included in the analysis.
  Participants
    Subfoveal | 39163
    Extrafoveal | 29400

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Acuity (VA) in Participant's Study Eye
Description: Change in visual acuity (VA) in participant's study eye is reported. Study eye is defined as the first eye with the disease, and fellow eye, the participant's second eye. Change in VA was determined by calculating the difference between mean visual acuity (VA) readings at index diagnosis, and mean at another timepoint, assessed yearly for participants with valid VA readings at both timepoints.
Time Frame: From index date of GA diagnosis up to 5 years
Population: Participants with GA at the index date and at least one year of follow-up data, with a VA reading at index, and at least one more VA reading at a subsequent follow-up year. The populations were different for each year since patients should have certain follow-up information to contribute to each cohort, and some participants had data in more than one year. Only those participants with VA readings at appropriate timepoints, with appropriate follow up, were analyzed.
Measure: Mean (95% Confidence Interval); unit: Letters read
Groups:
- Patients With Geographic Atrophy (GA): Patients diagnosed with geographic atrophy (GA) in at least one eye, at least 50 years old, with information on laterality and registered in the Vestrum health database between January 2015 and April 2023.
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 25477
Letters read
  Change in VA (Year 1): number analyzed (Participants) | 18455
  Change in VA (Year 1) | -2.8 [-3.0 to -2.6]
  Change in VA (Year 2): number analyzed (Participants) | 14856
  Change in VA (Year 2) | -5.9 [-6.2 to -5.6]
  Change in VA (Year 3): number analyzed (Participants) | 9485
  Change in VA (Year 3) | -8.6 [-9.0 to -8.2]
  Change in VA (Year 4): number analyzed (Participants) | 6304
  Change in VA (Year 4) | -10.3 [-10.9 to -9.8]
  Change in VA (Year 5): number analyzed (Participants) | 3809
  Change in VA (Year 5) | -11.9 [-12.6 to -11.2]

2. Primary Outcome: Number of Participants Who Developed or Progressed to Age-related Macular Degeneration (wAMD) in the Study Eye
Description: Number of participants who developed or progressed to age-related macular degeneration (wAMD) in the study eye is reported. The criteria used to determine progression through development to wAMD was identifying when ICD (International Classification of Diseases) codes for wAMD were present in the study eye.
Time Frame: From index date of GA diagnosis up to 5 years.
Population: Participants with GA at the index date and at least one year of follow-up data, excluding patients with wAMD prior to index. Only participants with appropriate follow up were analyzed. The populations were different for each year since patients should have certain follow-up information to contribute to each cohort, and some participants had data in more than one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 27974
Participants
  Participants with wAMD in 1+ years | 1866
  Participants with wAMD in 2+ years: number analyzed (Participants) | 18673
  Participants with wAMD in 2+ years | 2271
  Participants with wAMD in 3+ years: number analyzed (Participants) | 12552
  Participants with wAMD in 3+ years | 2191
  Participants with wAMD in 4+ years: number analyzed (Participants) | 8080
  Participants with wAMD in 4+ years | 1764
  Participants with wAMD in 5+ years: number analyzed (Participants) | 4743
  Participants with wAMD in 5+ years | 1247

3. Primary Outcome: Number of Participants Who Developed or Progressed to Geographic Atrophy (GA) in the Fellow Eye
Description: Number of participants who developed or progressed to geographic atrophy (GA) in the fellow eye is reported. For patients diagnosed with GA at baseline, the development of GA in the fellow eye was closely monitored over time, with progress tracked for each year.
Time Frame: From index date of GA diagnosis up to 5 years.
Population: Participants with GA at the index date and at least one year of follow-up data, excluding bilateral patients at index. Only participants with appropriate follow up were analyzed. The populations were different for each year since patients should have certain follow-up information to contribute to each cohort, and some participants had data in more than one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 19946
Participants
  Participants with GA in fellow eye in 1+ years | 1102
  Participants with GA in fellow eye in 2+ years: number analyzed (Participants) | 13626
  Participants with GA in fellow eye in 2+ years | 1319
  Participants with GA in fellow eye in 3+ years: number analyzed (Participants) | 9278
  Participants with GA in fellow eye in 3+ years | 1207
  Participants with GA in fellow eye in 4+ years: number analyzed (Participants) | 6060
  Participants with GA in fellow eye in 4+ years | 936
  Participants with GA in fellow eye in 5+ years: number analyzed (Participants) | 3654
  Participants with GA in fellow eye in 5+ years | 635

4. Primary Outcome: Change in Lesion Location for Participants With wAMD in Study Eye
Description: Change in lesion location from extrafoveal to subfoveal in participants who developed wAMD in study eye is reported. Lesion location was assessed at index diagnosis and at each year, then stratified by whether a patient developed wAMD in the 5 years post diagnosis. Changes in lesion were calculated as the difference in the number of participants with extrafoveal location at index diagnosis of the study eye, compared to the number of participants with extrafoveal lesion in the study eye at each year.
Time Frame: From index date of GA diagnosis up to 5 years
Population: Participants with GA at index date and five years of follow-up data who developed wAMD in the study eye after the index date. The populations were different for each year since only patients with lesion location information contributed to each cohort. Only participants with appropriate follow up were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 3449
Participants
  Participants with change of lesion location in Year 1: number analyzed (Participants) | 1073
  Participants with change of lesion location in Year 1 | 9
  Participants with change of lesion location in Year 2: number analyzed (Participants) | 843
  Participants with change of lesion location in Year 2 | 26
  Participants with change of lesion location in Year 3: number analyzed (Participants) | 636
  Participants with change of lesion location in Year 3 | 28
  Participants with change of lesion location in Year 4: number analyzed (Participants) | 496
  Participants with change of lesion location in Year 4 | 31
  Participants with change of lesion location in Year 5: number analyzed (Participants) | 401
  Participants with change of lesion location in Year 5 | 44

5. Primary Outcome: Change in Lesion Location for Participants With GA in Fellow Eye
Description: Change in lesion location from extrafoveal to subfoveal in participants who developed GA in fellow eye is reported. Lesion location was assessed at index diagnosis and at each year, then stratified by whether a patient developed GA in the 5 years post diagnosis. Changes in lesion were calculated as the difference in the number of participants with extrafoveal location at index diagnosis of the study eye, compared to the number of participants with extrafoveal lesion in the study eye at each year.
Time Frame: From index date of GA diagnosis up to 5 years
Population: Participants with GA at the index date and five years of follow-up data who developed GA in the fellow eye after the index date. The populations were different for each year since only patients with lesion location information contributed to each cohort. Only participants with appropriate follow up were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 2671
Participants
  Participants with change of lesion location in Year 1: number analyzed (Participants) | 579
  Participants with change of lesion location in Year 1 | 27
  Participants with change of lesion location in Year 2: number analyzed (Participants) | 535
  Participants with change of lesion location in Year 2 | 41
  Participants with change of lesion location in Year 3: number analyzed (Participants) | 522
  Participants with change of lesion location in Year 3 | 59
  Participants with change of lesion location in Year 4: number analyzed (Participants) | 509
  Participants with change of lesion location in Year 4 | 67
  Participants with change of lesion location in Year 5: number analyzed (Participants) | 526
  Participants with change of lesion location in Year 5 | 89

6. Primary Outcome: Occurrence of GA Over Study Period
Description: Incidence and prevalence of GA over time is reported. This endpoint analyzed the yearly counts of newly diagnosed or prevalent cases to help in understanding the progression of the overall disease.
Time Frame: Number of yearly counts of GA from 2018 to 2013, by quarterly average.
Population: Participants newly diagnosed with GA by quarterly average per year, for 2018-2023. Given the nature of the database, it was not possible to assess the prevalence or incidence of GA, but the absolute numbers of first time GA diagnosis, which is presented here.
Measure: Number; unit: Number of participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 48832
Number of participants
  Total new diagnosis of GA patients by quarterly average in 2018 | 2208
  Total new diagnosis of GA patients by quarterly average in 2019 | 2227
  Total new diagnosis of GA patients by quarterly average in 2020 | 1881
  Total new diagnosis of GA patients by quarterly average in 2021 | 2273
  Total new diagnosis of GA patients by quarterly average in 2022 | 2388
  Total new diagnosis of GA patients by quarterly average in 2023 | 3307

7. Secondary Outcome: Retinal Disease-related Outcomes: Number of Visits Per Quarter in a Year
Description: The retinal disease-related healthcare resource utilization (HCRU) outcome, number of visits by participants per quarter in a year is reported.
Time Frame: Mean number of quarterly visits from 2019 up to 2023.
Population: Participants were evaluated from the incident date of GA and assessed on a yearly basis for changes in physician habits over time. A patient visit or encounter was identified in the database any time a patient visited one of the panel physicians, without filtering on follow-up information. Results are presented only for first quarters of 2019 to 2023 respectively.
Measure: Mean (Standard Deviation); unit: Mean number of visits per quarter
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 68563
Mean number of visits per quarter
  Mean number of visits in first quarter of 2019: number analyzed (Participants) | 20231
  Mean number of visits in first quarter of 2019 | 0.990 (0.97)
  Mean number of visits in first quarter of 2020: number analyzed (Participants) | 21749
  Mean number of visits in first quarter of 2020 | 0.983 (0.99)
  Mean number of visits in first quarter of 2021: number analyzed (Participants) | 23045
  Mean number of visits in first quarter of 2021 | 1.032 (1.01)
  Mean number of visits in first quarter of 2022: number analyzed (Participants) | 24280
  Mean number of visits in first quarter of 2022 | 1.057 (0.99)
  Mean number of visits in first quarter of 2023: number analyzed (Participants) | 21648
  Mean number of visits in first quarter of 2023 | 1.373 (0.90)

8. Secondary Outcome: Retinal Disease-related Outcomes: Number of Anti-VEGF Injections Per Quarter
Description: The retinal disease-related healthcare resource utilization (HCRU) outcome, number of anti-vascular endothelial growth factor (anti-VEGF) injections per quarter in a year is reported.
Time Frame: Mean number of quarterly anti-VEGF injections from 2019 up to 2023.
Population: Participants were evaluated from index diagnosis and last encounter date, including patients in quarters with no anti-VEGF treatments, without filtering on follow-up information. Results are presented only for first quarters of 2019 to 2023 respectively.
Measure: Mean (Standard Deviation); unit: Mean number of anti-VEGF injections
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 68563
Mean number of anti-VEGF injections
  Mean number of anti-VEGF injections in first quarter of 2019: number analyzed (Participants) | 20231
  Mean number of anti-VEGF injections in first quarter of 2019 | 0.233 (0.63)
  Mean number of anti-VEGF injections in first quarter of 2020: number analyzed (Participants) | 21749
  Mean number of anti-VEGF injections in first quarter of 2020 | 0.250 (0.65)
  Mean number of anti-VEGF injections in first quarter of 2021: number analyzed (Participants) | 23045
  Mean number of anti-VEGF injections in first quarter of 2021 | 0.275 (0.68)
  Mean number of anti-VEGF injections in first quarter of 2022: number analyzed (Participants) | 24280
  Mean number of anti-VEGF injections in first quarter of 2022 | 0.295 (0.70)
  Mean number of anti-VEGF injections in first quarter of 2023: number analyzed (Participants) | 21648
  Mean number of anti-VEGF injections in first quarter of 2023 | 0.442 (0.82)

9. Secondary Outcome: Retinal Disease-related Outcomes: Number of Participants With Ocular Comorbidities by Year of Follow up
Description: The retinal disease-related HCRU outcome, number of ocular comorbidities by year of follow up is reported.
Time Frame: Total number of participants with ocular comorbidities were documented from index date up to 5 years.
Population: Participants with GA were tracked longitudinally (yearly) from index date of GA diagnosis in the database for occurrence of ocular comorbidities.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 68563
Participants
  Participants with ocular comorbidities in study eye: on or before index | 36518
  Participants with ocular comorbidities in study eye: in the first year | 38507
  Participants with ocular comorbidities in study eye: in the first 2 years | 39506
  Participants with ocular comorbidities in study eye: in the first 3 years | 40077
  Participants with ocular comorbidities in study eye: in the first 4 years | 40382
  Participants with ocular comorbidities in study eye: in the first 5 years | 40546

10. Secondary Outcome: HCRU Outcome: Number of Participants With the Medical Procedure of Corneal Transplant
Description: The number of participants with corneal transplant during the observational period is reported.
Time Frame: Total number of participants with corneal transplants were documented from index date up to 5 years.
Population: Participants with GA were tracked longitudinally (yearly) from index date of GA diagnosis in the database for occurrence of corneal transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 68563
Participants
  Participants with corneal transplant in study eye: on or before index | 6
  Participants with corneal transplant in study eye: in the first year | 7
  Participants with corneal transplant in study eye: in the first 2 years | 8
  Participants with corneal transplant in study eye: In the first 3 years | 10
  Participants with corneal transplant in study eye: in the first 4 years | 11
  Participants with corneal transplant in study eye: in the first 5 years | 11

11. Secondary Outcome: HCRU Outcome: Number of Participants With the Medical Procedure of Incisional Glaucoma Surgery
Description: Number of participants with incisional glaucoma surgery during the observational period is reported.
Time Frame: Total number of participants with incisional glaucoma surgery were documented from index date up to 5 years.
Population: Participants with GA were tracked longitudinally (yearly) from index date of GA diagnosis in the database for occurrence of incisional glaucoma surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 68563
Participants
  Participants with incisional glaucoma surgery in study eye: on or before index | 0
  Participants with incisional glaucoma surgery in study eye: in the first year | 0
  Participants with incisional glaucoma surgery in study eye: in the first 2 years | 0
  Participants with incisional glaucoma surgery in study eye: in the first 3 years | 0
  Participants with incisional glaucoma surgery in study eye: in the first 4 years | 0
  Participants with incisional glaucoma surgery in study eye: in the first 5 years | 0

12. Secondary Outcome: HCRU Outcome: Number of Participants With the Medical Procedure of Vitrectomy
Description: Number of participants with vitrectomy during the observational period is reported.
Time Frame: Total number of participants with vitrectomy were documented from index date up to 5 years.
Population: Participants with GA were tracked longitudinally (yearly) from index date of GA diagnosis in the database for occurrence of vitrectomy.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Geographic Atrophy (GA)
Number analyzed (Participants) | 68563
Participants
  Participants with vitrectomy performed on study eye: on or before index | 1579
  Participants with vitrectomy performed on study eye: in the first year | 1858
  Participants with vitrectomy performed on study eye: in the first 2 years | 1955
  Participants with vitrectomy performed on study eye: in the first 3 years | 1995
  Participants with vitrectomy performed on study eye: in the first 4 years | 2038
  Participants with vitrectomy performed on study eye: in the first 5 years | 2062

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: This was an observational study using existing electronic health care records with data retrieved from the Vestrum Health database in the US.
  No adverse events were collected on an individual case level as no safety reporting was applicable for the study.
Arm/Group | Patients With Geographic Atrophy (GA)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The Vestrum database used in this study included only data from visits that occurred at the practices contributing to the database, therefore anything occurring during visits to a retinal specialist in a different practice, state, country etc. was not captured. An overall limitation of the dataset is that data is typically entered by the physician, therefore there is no real-time validation of the information entered during the encounter either in terms of completeness or accuracy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT05891275/Prot_SAP_000.pdf